CLINICAL TRIAL: NCT05085782
Title: Reconsolidation Therapy With Propranolol as a Novel Treatment for Chronic Pain : a Placebo-controlled Feasibility Study
Brief Title: Reconsolidation Therapy With Propranolol as a Treatment for Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-4092
Record Dates: First submitted 2021-09-27; First posted 2021-10-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low-back Pain; Fibromyalgia
Keywords: Chronic pain; Reconsolidation therapy; Propranolol; Treatment
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Propranolol; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): 1. Pain neuroscience education (10 short videos - 2 to 4 mins each)
  2. 6 weekly sessions of Reconsolidation therapy with propranolol. At the beginning of each session, participants will take 2 to 4 capsules of 20 mg propranolol (dose calculated based on sex and height). One hour after ingestion of the propranolol, participants will undergo a reactivation procedure, wherein they will be asked to describe/visualize painful movements/activities.
  Interventions: Drug: Propranolol Hydrochloride; Behavioral: Reactivation procedure; Behavioral: Pain neuroscience education
- Placebo (Placebo Comparator): 1. Pain neuroscience education (10 short videos - 2 to 4 mins each)
  2. 6 weekly sessions of Reconsolidation therapy with a placebo. At the beginning of each session, participants will take 2 to 4 capsules of 20 mg placebo (dose calculated based on sex and height). One hour after ingestion of the placebo, participants will undergo a reactivation procedure, wherein they will be asked to describe/visualize painful movements/activities.
  Interventions: Drug: Placebo; Behavioral: Reactivation procedure; Behavioral: Pain neuroscience education

INTERVENTIONS:
Drug: Propranolol Hydrochloride — 6 weekly doses (40 to 80 mg) 1h before the reactivation procedure
  Other Names: Experimental group
  Arms: Propranolol
Drug: Placebo — 6 weekly doses (40 to 80 mg) 1h before the reactivation procedure
  Other Names: Control group
  Arms: Placebo
Behavioral: Reactivation procedure — Description/visualization of painful movements/activities
Behavioral: Pain neuroscience education — In the form of 10 videos that participants will watch on their own time

SUMMARY:
The primary aim of this study is to document the feasibility and acceptability of an intervention consisting of pain neuroscience education and reconsolidation therapy with propranolol in adults suffering from chronic pain (chronic low back pain or fibromyalgia).

The secondary aim of the study is to estimate the effect size of the intervention on pain and function one month post-intervention, and to obtain data for sample-size calculation for a subsequent randomized controlled trial.

DETAILED DESCRIPTION:
Background: Many patients with chronic pain exhibit abnormal synaptic changes in the central nervous system - including hyperactivity in the amygdala - reminiscent of those seen in post-traumatic stress disorder (PTSD). A recently developed psychiatric treatment for PTSD involves reactivating the synapses to make them temporarily malleable and then blocking their reconsolidation with propranolol, thereby reducing the hyperactivity in the amygdala and decreasing the intensity of the symptoms in a lasting way. Considering the similarities between PTSD and chronic pain, this treatment could also be beneficial for patients with chronic pain.

Objectives: The primary objective of this study will be to document the feasibility and acceptability of a combined pain neuroscience education and reconsolidation blockade intervention with oral propranolol (or placebo) in adult patients with chronic pain (specifically, low back pain or fibromyalgia). The secondary objective will be to estimate the effect size of the intervention on function and pain one month post-intervention, and to obtain the data necessary for a sample size calculation of a subsequent larger scale study.

Description: The research design is a quantitative, placebo-controlled clinical trial (Phase II) feasibility study. The sample will consist of French-speaking adults with chronic low back pain or fibromyalgia (n=24 per population; 12 control and 12 experimental participants for each population; allocation by minimization); participants with a contraindication to propranolol or a neurological diagnosis will be excluded. All participants will receive education on the neuroscience of pain (video vignettes) and will participate in 6 weekly intervention sessions. During these sessions, they will receive propranolol or placebo capsules (double-blind; dosing based on size) and participate in a reactivation procedure (description and/or visualization of painful movements). Feasibility measures will be collected throughout the study; acceptability and efficacy measures will be assessed 4 weeks post-intervention, with the exception of physical function (primary efficacy measure), which will also be measured at each intervention session.

Relevance: This study will be the first to use reconsolidation blockade for the treatment of chronic pain. The postulated mechanism of action is plausible and supported by scientific evidence, but to date has never been tested in humans with persistent pain. If our results demonstrate that the intervention is feasible, acceptable, and has the potential to be effective, randomized clinical trials may follow our study to robustly evaluate the effect of our intervention in the short and long term. The intervention could also be evaluated in other chronic pain populations with central sensitization, such as pelvic pain, chronic neck pain (whiplash), etc.

ELIGIBILITY:
Inclusion Criteria:

* French speaking
* Suffering from [chronic low back pain OR fibromyalgia] for >6 months
* Average pain at least 4/10
* Central sensitization (assessed via a standardized physiotherapy evaluation and the Central Sensitization Inventory)

Exclusion Criteria:

* Health condition for which propranolol is contra-indicated
* Medication with which co-administration of propranolol is contra-indicated
* Severe or uncontrolled neurological/psychiatric condition (including post-traumatic stress disorder, substance abuse, suicidal ideation, etc.)
* Surgery of the lower-back in the last 3 years
* Litigation surrounding the painful condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome 1 : Weekly recruitment rate | Through recruitment phase (estimated 3 months per population)
  Number of prospective participants successfully recruited every week, vs number of participants excluded and number of refusals
Feasibility outcome 2 : Rate of study completion | Through data collection phase (estimated 6 months per population)
  Percentage of sample with perfect attendance vs partial attendance vs withdrawal vs exclusion vs loss to follow-up.
Feasibility outcome 3 : Number of participants with adverse events (observed and self-reported) | Through data collection phase (estimated 6 months per population)
  For all adverse even, the following will be reported : Type & severity (according to the CTCAE), attribution, expected vs unexpected
Feasibility outcome 4 : % participants in each group who believe they received the experimental treatment (propranolol) | At follow-up (on average,12 weeks after recruitment)
  This percentage will be compared between the two groups to assess blinding
Acceptability outcome 1 : perceived burden of the intervention (prospective and retrospective) | Prospective rating : at baseline ; Retrospective rating : at follow-up (on average,12 weeks after recruitment)
  Rated on an 11-point numerical rating scale (0-10; 10 = worse outcome)
Acceptability outcome 2 : perceived ethicality of the intervention (prospective and retrospective) | Prospective rating : at baseline ; Retrospective rating : at follow-up (on average,12 weeks after recruitment)
  Rated on an 11-point numerical rating scale (0-10; 10 = better outcome)
Acceptability outcome 3 : perceived coherence of the intervention (prospective and retrospective) | Prospective rating : at baseline ; Retrospective rating : at follow-up (on average,12 weeks after recruitment)
  Rated on an 11-point numerical rating scale (0-10; 10 = better outcome)
Acceptability outcome 4 : perceived effectiveness of the intervention (prospective and retrospective) | Prospective rating : at baseline ; Retrospective rating : at follow-up (on average,12 weeks after recruitment)
  Rated on an 11-point numerical rating scale (0-10; 10 = better outcome)
Acceptability outcome 5 : perceived self-efficacy relating to the intervention (prospective and retrospective) | Prospective rating : at baseline ; Retrospective rating : at follow-up (on average,12 weeks after recruitment)
  Rated on an 11-point numerical rating scale (0-10; 10 = better outcome)

SECONDARY OUTCOMES:
Change in Physical functioning | From baseline to follow-up (approx 12 weeks)
  Measured using the self-reported Brief pain inventory (short form); (0-70; 70 = worse outcome)
Change in Pain intensity | From baseline to follow-up (approx 12 weeks)
  Measured using the self-reported Brief pain inventory (short form) (0-40; 40 = worse outcome)
Change in Emotional functioning | From baseline to follow-up (on average, 12 weeks)
  Measured using the self-reported Profile of mood states (-32 to 200; 200 = worse outcome)
Change in Central sensitization | From baseline to follow-up (on average, 12 weeks)
  Measured using the self-reported Central sensitization inventory (0-100; 100=worse outcome)
Change in Symptoms of fibromyalgia | From baseline to follow-up (on average, 12 weeks)
  Measured using the self-reported Fibromyalgia impact questionnaire(for the fibromyalgia population only) (0=100; 100 = worse outcome)
Participant ratings of global improvement and satisfaction with treatment | Follow-up (on average, 12 weeks after recruitment)
  Measured using the self-reported Patient global impression of change (1-7; 7 = better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Leonard, PhD, Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Centre de recherche sur le vieillissement (CdRV), Sherbrooke, Quebec
  - CRCHUS: Centre de recherche du centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No